CLINICAL TRIAL: NCT04455620
Title: Phase I/IIa, First-in-human, Open-label, Dose Escalation Trial With Expansion Cohorts to Evaluate Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of BNT151 as a Monotherapy and in Combination With Other Anti-cancer Agents in Patients With Solid Tumors
Brief Title: BNT151 as a Monotherapy and in Combination With Other Anti-cancer Agents in Patients With Solid Tumors
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT151-01; 2019-003572-39 (EudraCT Number)
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor
Keywords: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1: BNT151 (Experimental): Monotherapy dose escalation in participants with advanced solid malignancies until the MTD and/or RP2D
  Interventions: Biological: BNT151

INTERVENTIONS:
Biological: BNT151 — intravenous (IV)

SUMMARY:
This was an open-label, multicenter Phase I/IIa dose escalation, safety, pharmacokinetic and pharmacodynamic (PD) study of BNT151 with expansion cohorts in various solid tumor indications.

The study was planned to be performed in Part 1, Part 2A, and Part 2B with adaptive design elements. Part 2 was not conducted because of the clinical study being terminated early.

The monotherapy dose escalation, (Part 1) of this clinical study enrolled participants with various solid tumors that are metastatic or of advanced unresectable stage for whom there was no available standard therapy likely to confer clinical benefit, or participants who are not candidates for such available therapy. Dose escalation followed an accelerated titration design, i.e., started with single participant cohorts followed by larger participant cohorts informed by the 3+3 design.

Part 1 of the study also planed to implement a dedicated biomarker cohort in BNT151 monotherapy. The biomarker cohort was planned to recruit participants at selected sites in the United States (US) only. The objective of the cohort was to observe PD activity and drug-induced changes in the blood and tumor and only to generate data for exploratory endpoints or additional research. However, the biomarker cohort was not opened, and therefore no data were generated.

During combination dose escalation (Part 2A), participants with squamous cell carcinoma of head and neck, and hepatocellular carcinoma were planned to be enrolled and treated with a combination of BNT151 and pembrolizumab. Once Part 2A was completed, participants with renal cell carcinoma, non-small cell lung cancer, and triple negative breast cancer were planned to be enrolled (Part 2B) and treated with a combination of BNT151 with the respective standard of care (SoC).

DETAILED DESCRIPTION:
The study was terminated early due to sponsor's decision after careful considerations including recruitment projections and available data, and not due to any safety concerns. At the time of the termination, fewer dose levels were tested than anticipated.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histological documentation of the original primary tumor via a pathology report.
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

For Part 1:

* Histologically confirmed solid tumor that is metastatic or of advanced unresectable stage and for whom there is no available standard therapy likely to confer clinical benefit, or participant who is not a candidate for such available therapy. If there is no contraindication, participants should have exhausted all SoC therapies before entering the study, if possible.

For all Parts:

* ≥18 years of age.
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose and procedures required for the study and are willing to participate in the study prior to any study-related assessments or procedures.
* Eastern Cooperative Oncology Group performance status of 0 to 1.
* Adequate coagulation function at screening as required by the protocol.
* Adequate hematologic function at screening as required by the protocol.
* Adequate hepatic function at screening as required by the protocol.
* Adequate renal function at screening as required by the protocol.
* Able and willing to attend study visits as required by the protocol.
* Women of childbearing potential (WOCBP) must have a negative serum (beta-human chorionic gonadotropin) test/value at screening. Participants who are postmenopausal or permanently sterilized can be considered as not having reproductive potential.
* WOCBP must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire study, until 6 months after last BNT151 treatment.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control, e.g. either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 6 months after receiving the last dose of BNT151.
* WOCBP must agree to use highly effective contraception during the study and for 6 months after receiving the last dose of BNT151. Birth control methods are considered highly effective if they have a failure rate of less than 1% per year, when used consistently and correctly.
* Biomarker cohort: At selected US sites only: at enrollment participants must agree to have one pre-dose biopsy and lesion that is deemed accessible by the investigator. If possible, at least one on-treatment biopsy should be accessible from same tumor lesion.

EXCLUSION CRITERIA:

* Use of any investigational medical product (IMP) or device within 28 days before administration of first dose of study treatment.
* Has been receiving: radiotherapy, chemotherapy, or molecularly-targeted agents or tyrosine kinase inhibitors within 2 weeks or 5 half-lives (whichever is longer) of the start of study treatment; immunotherapy/monoclonal antibodies within 3 weeks of the start of study treatment; any live vaccine within 4 weeks of the start of study treatment; nitrosoureas, antibody-drug conjugates, or radioactive isotopes within 6 weeks of the start of study treatment.
* Ongoing participation in the active treatment phase of interventional clinical study.
* Receives concurrent systemic (oral or IV) steroid therapy >10 mg prednisone daily or its equivalent for an underlying condition.
* Has had major surgery within the 4 weeks before the first dose of BNT151.
* Ongoing or active infection requiring IV treatment with anti-infective therapy that has been administered less than 2 weeks prior to the first dose of BNT151.
* Has ongoing side effects to any prior therapy or procedures for any medical condition not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0 Grade ≤1.

Medical conditions:

* Current evidence of new or growing brain or leptomeningeal metastases during screening. Participants with known brain metastases may be eligible if they:
* had radiotherapy, surgery or stereotactic surgery for the brain metastases;
* have no neurological symptoms (excluding Grade ≤2 neuropathy);
* have stable brain metastasis on the computed tomography or magnetic resonance imaging scan within 4 weeks before signing the informed consent;
* are not undergoing acute corticosteroid therapy or steroid taper.
* Has a history of a cerebrovascular accident or transient ischemic attack less than 6 months ago.
* Effusions (pleural, pericardial, or ascites) requiring drainage.
* History of autoimmune disease active or past including but not limited to inflammatory bowel disease, systemic lupus erythematosus, ankylosing spondylitis, scleroderma, or multiple sclerosis. Has any active immunologic disorder requiring immunosuppression with steroids or other immunosuppressive agents (e.g., azathioprine, cyclosporine A) with the exception of participants with isolated vitiligo, resolved childhood asthma or atopic dermatitis, controlled hypoadrenalism or hypopituitarism, and participants with a history of Grave's disease with stable thyroid function. Participants with controlled hyperthyroidism must be negative for thyroglobulin, thyroid peroxidase antibodies, and thyroid stimulating immunoglobulin prior to administration of study treatment.
* Known history of seropositivity for human immunodeficiency virus (HIV) with CD4+ T-cell (CD4+) counts <350 cells/µL and with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections.
* Known history/positive serology for hepatitis B requiring active antiviral therapy (unless immune due to vaccination or resolved natural infection or unless passive immunization due to immunoglobulin therapy). Participants with positive serology must have hepatitis B viral load below the limit of quantification.
* Active hepatitis C virus (HCV) infection; participants who have completed curative antiviral treatment with HCV viral load below the limit of quantification are allowed.
* Any contraindication to the combination therapies as per United States Prescribing Information or Summary of Product Characteristics for participants receiving BNT151 in combination with other systemic anticancer agent(s).
* Another primary malignancy that has not been in remission for at least 2 years, with the exception of those with a negligible risk of metastasis or death (including but not limited to adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ).

Other comorbidities:

* Abnormal electrocardiograms that are clinically significant, such as Fridericia-corrected QT prolongation >480 ms.
* In the opinion of the treating investigator, has any concurrent conditions that could pose an undue medical hazard or interfere with the interpretation of the study results; these conditions include, but are not limited to:
* Ongoing or active infection requiring antibiotic/antiviral/antifungal therapy
* Concurrent congestive heart failure (New York Heart Association Functional Classification Class III or IV)
* Concurrent unstable angina
* Concurrent cardiac arrhythmia requiring treatment (excluding asymptomatic atrial fibrillation)
* Acute coronary syndrome within the previous 6 months
* Pulmonary embolism within the previous 3 months
* Significant pulmonary disease (shortness of breath at rest or on mild exertion) for example due concurrent severe obstructive pulmonary disease.
* Cognitive, psychological or psychosocial impediment that would impair the ability of the participant to receive therapy according to the protocol or adversely affect the ability of the participant to comply with the informed consent process, protocol, or protocol-required visits and procedures.
* Is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2024-05-28 (Actual); Study Completion 2024-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (6):
- United States (4):
  - Yale Cancer Center, New Haven, Connecticut
  - Sarah Cannon Research Institute at Tennessee Oncology, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Spain (2):
  - Vall d´Hebron Institute of Oncology (VHIO), Barcelona
  - START Madrid - HM CIOCC, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at centers experienced in first-in-human studies in two countries, i.e., the US and Spain.
Pre-assignment Details: A total of 49 participants were enrolled in this study and all participants received at least one dose of the IMP.
Groups:
- BNT151 0.4 ug/kg; BNT151 2.0 ug/kg; BNT151 4.0 ug/kg; BNT151 8.0 ug/kg: Participants from Part 1 treated with BNT151 monotherapy. BNT151 was administered intravenously on Day 1 of each 3-week treatment cycle (Q3W; 21 days).
- BNT151 2.0 + 4.0 ug/kg: Participants from Part 1 treated with BNT151 monotherapy with pre-conditioning. Treatment started with a pre-conditioning dose (a lower dose of 2 μg/kg) on Day 1 of the pre-conditioning cycle (cycle of 7 days). The participants then received the intended dose of 4 μg/kg at the discretion of the safety review committee (SRC) on Day 1 of every Q3W treatment cycle.
Period: Overall Study
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Started | 1 | 8 | 24 | 2 | 14
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 8 | 24 | 2 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 0
Not completed — Death | 1 | 6 | 20 | 1 | 7
Not completed — Study Termination | 0 | 2 | 1 | 0 | 6

BASELINE CHARACTERISTICS:
Population: Treated set, i.e., defined as all participants who received IMP (i.e., at least one dose of BNT151).
Groups:
- BNT151 2.0 + 4.0 ug/kg: Participants from Part 1 treated with BNT151 monotherapy with pre-conditioning. Treatment started with a pre-conditioning dose (a lower dose of 2 μg/kg) on Day 1 of the pre-conditioning cycle (cycle of 7 days). The participants then received the intended dose of 4 μg/kg at the discretion of the SRC on Day 1 of every Q3W treatment cycle.
- Total: Total of all reporting groups
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg | Total
Number analyzed (Participants) | 1 | 8 | 24 | 2 | 14 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 7 | 13 | 1 | 6 | 27
  >=65 years | 1 | 1 | 11 | 1 | 8 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 9 | 1 | 8 | 22
  Male | 1 | 4 | 15 | 1 | 6 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 5 | 0 | 3 | 9
  Not Hispanic or Latino | 1 | 5 | 15 | 1 | 6 | 28
  Unknown or Not Reported | 0 | 2 | 4 | 1 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 0 | 2
  White | 1 | 7 | 18 | 2 | 7 | 35
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 5 | 0 | 6 | 11
Body mass index (BMI) category [Number; unit: participants]
  <18 kg/m^2 | 0 | 0 | 0 | 0 | 1 | 1
  ≥18 to <25 kg/m^2 | 0 | 2 | 8 | 0 | 6 | 16
  ≥25 to <30 kg/m^2 | 0 | 2 | 8 | 1 | 6 | 17
  ≥30 kg/m^2 | 1 | 4 | 8 | 1 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) During the DLT Evaluation Period in Part 1
Time Frame: From first dose of IMP up to 21 days (Cycle 1).
Population: DLT evaluable set, including all participants from the safety set who were enrolled in dose-escalation cohorts and either experienced a DLT during the DLT evaluation period (Cycle 1) or completed the DLT evaluation period.
  Participants who did not experience any DLT during the DLT observation period were considered to be evaluable if they have been observed for minimum 21 days following the first dose and were considered to have sufficient safety data to conclude that a DLT did not occur.
Measure: Number; unit: participants
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Number analyzed (Participants) | 1 | 8 | 24 | 2 | 14
participants | 0 | 0 | 0 | 2 | 0

2. Primary Outcome: Number of Participants With at Least One Treatment Emergent Adverse Event (TEAE) Including Grade ≥3, Serious, Fatal TEAE by Relationship
Description: A TEAE was defined as any adverse event (AE) with an onset date on or after the first administration of IMP (if the AE was absent before the first administration of IMP) or worsened after the first administration of IMP (if the AE was present before the first administration of IMP). AEs with an onset date more than 60 days after the last administration of IMP were considered as treatment emergent only if assessed as related to IMP by the investigator.
  The intensity of an TEAE was graded according to the NCI CTCAE version 5.0. Grade 3=Severe, Grade 4=Life threatening, Grade 5=Death.
Time Frame: From first dose of IMP through study completion, a maximum of 30 months.
Population: Safety set, i.e., all participants who received IMP (i.e., at least one dose of BNT151).
Measure: Count of Participants; unit: Participants
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Number analyzed (Participants) | 1 | 8 | 24 | 2 | 14
Participants
  TEAE | 1 | 8 | 24 | 2 | 14
  TEAE related to BNT151 | 0 | 7 | 23 | 2 | 11
  Grade ≥3 TEAE | 1 | 3 | 14 | 2 | 5
  Grade ≥3 TEAE related to BNT151 | 0 | 3 | 8 | 1 | 2
  TEAE related to study procedure | 0 | 0 | 0 | 0 | 2
  Serious TEAE | 0 | 3 | 9 | 2 | 4
  Serious TEAE related to BNT151 | 0 | 1 | 5 | 2 | 0
  Serious TEAE leading to death | 0 | 0 | 0 | 1 | 0
  Serious TEAE related to BNT151 leading to death | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Paticipants With at Least One TEAE Leading to Dose Reduction, Dose Interruption, and Treatment Discontinuation of BNT151
Description: A TEAE was defined as any AE with an onset date on or after the first administration of IMP (if the AE was absent before the first administration of IMP) or worsened after the first administration of IMP (if the AE was present before the first administration of IMP). AEs with an onset date more than 60 days after the last administration of IMP were considered as treatment emergent only if assessed as related to IMP by the investigator.
Time Frame: From first dose of IMP through treatment completion, a maximum of 24 months.
Population: Safety set, i.e., all participants who received IMP (i.e., at least one dose of BNT151).
Measure: Count of Participants; unit: Participants
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Number analyzed (Participants) | 1 | 8 | 24 | 2 | 14
Participants
  TEAE leading to dose reduction | 0 | 0 | 0 | 0 | 0
  TEAE leading to dose interruption | 0 | 0 | 4 | 0 | 2
  TEAE leading to permanent treatment discontinuation of BNT151 | 0 | 0 | 2 | 1 | 0

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants in whom a complete response (CR) or partial response (PR) (per RECIST version 1.1) was observed as best overall response.
  Confirmed ORR was defined as the proportion of participants in whom a CR or PR (per RECIST version 1.1) was observed as best overall response and has been confirmed with a subsequent assessment of objective response at least 4 weeks apart.
Time Frame: Through study completion, a maximum of 30 months.
Population: Treated set, i.e., defined as all participants who received IMP (i.e., at least one dose of BNT151).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Number analyzed (Participants) | 1 | 8 | 24 | 2 | 14
percentage of participants
  ORR | 0 [0.0 to 97.5] | 0 [0.0 to 36.9] | 4.2 [0.1 to 21.1] | 0 [0.0 to 84.2] | 7.1 [0.2 to 33.9]
  Confirmed ORR | 0 [0.0 to 97.5] | 0 [0.0 to 36.9] | 4.2 [0.1 to 21.1] | 0 [0.0 to 84.2] | 7.1 [0.2 to 33.9]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the proportion of participants in whom a CR or PR or stable disease (SD) (per RECIST version 1.1, SD assessed at least 6 weeks after first dose) was observed as best overall response.
Time Frame: Through study completion, a maximum of 30 months.
Population: Treated set, i.e., defined as all participants who received IMP (i.e., at least one dose of BNT151).
Measure: Number (95% Confidence Interval); unit: percentage of partients
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Number analyzed (Participants) | 1 | 8 | 24 | 2 | 14
percentage of partients | 0 [0 to 97.5] | 25 [3.2 to 65.1] | 25 [9.8 to 46.7] | 0 [0 to 84.2] | 42.9 [17.7 to 71.1]

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from first objective response (CR or PR per RECIST version 1.1) to first occurrence of objective tumor progression (progressive disease per RECIST version 1.1) or death from any cause, whichever occurred first.
  Reporting groups with zero participants with confirmed objective response are not included.
Time Frame: Through study completion, a maximum of 30 months.
Population: Treated set, i.e., defined as all participants who received IMP (i.e., at least one dose of BNT151).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | BNT151 4.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
Number analyzed (Participants) | 1 | 1
months | 6.5 [NA to NA] — Confidence interval values value could not be estimated. | NA [NA to NA] — Value could not be calculated because participant was censored as per SAP defined censoring rules (i.e., no progression / lost to follow up).

ADVERSE EVENTS:
Time Frame: Deaths and serious AEs: All events from the signing of the study-specific ICF until early study termination, i.e., up to 31 months. Other AEs: All TEAEs, i.e., AEs reported from the start of study drug treatment until until early study termination, i.e., up to 30 months.
Description: Other AEs: All TEAEs, i.e., any AE with an onset date on or after the first dose of BNT151 (if the AE was absent before the first dose) or worsened after the first dose of BNT151 (if the AE was present before the first dose). AEs with an onset date >60 days after the last dose of BNT151 were included only if assessed as related to BNT151 by the investigator.
  If a participant experienced more than one event in a category, the participant is counted only once in that category.
Arm/Group | BNT151 0.4 ug/kg | BNT151 2.0 ug/kg | BNT151 4.0 ug/kg | BNT151 8.0 ug/kg | BNT151 2.0 + 4.0 ug/kg
All-Cause Mortality (participants affected / at risk) | 1/1 | 6/8 | 20/24 | 1/2 | 7/14
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/8 | 9/24 | 2/2 | 4/14
Other Adverse Events (participants affected / at risk) | 1/1 | 8/8 | 24/24 | 2/2 | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT151 0.4 ug/kg (N=1) | BNT151 2.0 ug/kg (N=8) | BNT151 4.0 ug/kg (N=24) | BNT151 8.0 ug/kg (N=2) | BNT151 2.0 + 4.0 ug/kg (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 4 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BNT151 0.4 ug/kg (N=1) | BNT151 2.0 ug/kg (N=8) | BNT151 4.0 ug/kg (N=24) | BNT151 8.0 ug/kg (N=2) | BNT151 2.0 + 4.0 ug/kg (N=14)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 11 | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 1 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 5 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 5 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 7 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 4 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 3
Chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Chills (General disorders) | 0 | 1 | 3 | 0 | 3
Fatigue (General disorders) | 1 | 2 | 3 | 0 | 5
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 6 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 1 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 3 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 2 | 9 | 0 | 10
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 3 | 1 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 3 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 4 | 0 | 2
Lymphocyte count decreased (Investigations) | 1 | 4 | 12 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 1
Red blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 5 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Choluria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Embolism venous (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively study sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-12-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT04455620/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/20/NCT04455620/SAP_001.pdf